CLINICAL TRIAL: NCT05445375
Title: STrategic Education for Patients Undergoing PAD Surgery (STEPUP Clinical Trial)
Brief Title: STEPUP Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00215376
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current education regimen (No Intervention): Participants will be given a PAD pamphlet and ad hoc verbal teaching by vascular providers.
- Intervention (Active Comparator): Participants will be given the current education regimen and watch a 20 minute online PAD education video.
  Interventions: Other: PAD education video

INTERVENTIONS:
Other: PAD education video — 20-min online multi-media video
  Arms: Intervention

SUMMARY:
This study will test whether, among patients undergoing surgery for peripheral artery disease (PAD), the addition of an online multimedia patient education video to the current education regimen will improve PAD knowledge, activation, and self-care engagement. The study will randomize 150 participants to one of 2 groups: current education regimen vs. current education regiment with video. The primary outcome is stage of self-care engagement. Secondary outcomes are PAD knowledge, self-efficacy, and activation. A subset of participants will also be randomly selected to participate in semi-structured interviews. Study duration for participants is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing surgery for PAD in Division of Vascular Surgery at Northwestern Memorial Hospital

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete study protocol
* Previously viewed the PAD education video
* Participation in pilot study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Readiness to change self-care engagement | Baseline to six-month follow-up
  Change in readiness to change self-care behaviors will be compared between the 2 groups. Readiness to change self-care behavior will be assessed as 1 of 5 stages in the Transtheoretical Model. Change in readiness to change behavior will be calculated as the difference between stages at baseline and six month follow-up (direction and magnitude). Assessment will occur in paper survey.

SECONDARY OUTCOMES:
PAD knowledge and beliefs | Baseline to six-month follow-up
  Change in PAD knowledge and beliefs will be compared between the 2 groups. Knowledge and beliefs will be assessed using multiple-choice questions in a paper survey.
Self-efficacy | Baseline to six-month follow-up
  Change in self-efficacy will be compared between the 2 groups. Self-efficacy will be assessed using 5 questions adapted from the General Self-Efficacy Scale in a paper survey. Responses are recorded on a 5-point Likert scale. Summed scores will range from 5 (minimum, lowest level of self-efficacy) to 25 (maximum, highest level of self-efficacy). Change in self-efficacy will be calculated as the difference in sum scores.
Activation level | Baseline to six-month follow-up
  Change in activation level will be compared between the 2 groups. Activation level will be assessed using the 13-item Patient Activation Measure (PAM-13), a validated instrument, which will be administered in a paper survey. The activation score is based on a 0-100-point scale (0=minimum, 100=maximum).The activation score is can be used to segment individuals into one of 4 progressively higher levels of activation. Change in activation score and level will be calculated as a difference in PAM-13 scores and levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No